CLINICAL TRIAL: NCT07103031
Title: Targeting The Right Pediatric Migraine Patient: A Comorbidity-Oriented Approach To Propranolol Prophylaxis
Brief Title: Comorbidity-Based Propranolol Use in Pediatric Migraine
Status: Completed | Type: Observational
Sponsor: Kayseri University (Other)
Responsible Party: Principal Investigator, Özge BAYKAN ÇOPUROĞLU, Asst. Prof., Kayseri University
Other Study IDs: KayseriUniversity12; EC/IRB Number- 2021/12-14 (Other: Tepecik Training and Research Hospital)
Record Dates: First submitted 2025-07-14; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Migraine; Migraine Disorders, Brain; Vitamin D Deficiency
Keywords: Propranolol; Pediatric Migraine; Migraine Prophylaxis; Vitamin D Deficiency
MeSH Terms: conditions — Migraine Disorders; Vitamin D Deficiency | interventions — Behavior Therapy; Cognitive Behavioral Therapy; Propranolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Behavioral therapy group
  Interventions: Behavioral: Behavioral therapy
- Group 2: Propranolol group
  Interventions: Drug: Propranolol

INTERVENTIONS:
Behavioral: Behavioral therapy — Patients in PedMIDAS stage 1-2 (score ≤ 30) received behavioral therapy including lifestyle counseling, stress management techniques, sleep hygiene education, and individualized headache triggers review. Additionally, each patient was provided with a headache report card to self-monitor symptoms, triggers, and medication use over a 3-month period.
  Other Names: Cognitive-Behavioral Therapy
  Groups: Group 1
Drug: Propranolol — Patients in PedMIDAS stage 3-4 (score > 30) received oral propranolol treatment at a dose of 1-3 mg/kg/day, adjusted by weight and tolerance, for a total of 3 months. The medication was prescribed and monitored by a pediatric neurologist. Patients were followed with routine check-ups and adverse effects were recorded.
  Other Names: β-blocker
  Groups: Group 2

SUMMARY:
This observational retrospective cohort study aims to identify clinical and biochemical predictors of response to propranolol prophylaxis in pediatric migraine. A total of 178 children diagnosed with migraine between 2021 and 2023 were evaluated based on headache-related disability (PedMIDAS) and pain severity (VAS). Patients were treated either with behavioral therapy or propranolol (1-3 mg/kg/day) for 3 months.

DETAILED DESCRIPTION:
Migraine is a common and disabling neurological condition in the pediatric population, often requiring prophylactic treatment to reduce attack frequency and improve quality of life. Propranolol is frequently prescribed for pediatric migraine prevention; however, treatment response varies considerably among individuals. Understanding the clinical and biochemical factors that predict treatment efficacy could enhance individualized care and reduce unnecessary medication use.

This retrospective cohort study evaluated 178 children diagnosed with pediatric migraine between January 2021 and December 2023 at a tertiary neurology outpatient clinic. All participants were assessed using the Pediatric Migraine Disability Assessment Scale (PedMIDAS) and Visual Analog Scale (VAS) before and after treatment. Patients received either behavioral therapy or oral propranolol (1-3 mg/kg/day) for a duration of 3 months, based on clinical indication and family preference.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-20 years
* Diagnosed with primary headache according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)
* Clinical and/or neurological evaluation consistent with primary headache
* Completed baseline PedMIDAS and VAS assessments
* Available for 3-month follow-up after initiation of treatment

Exclusion Criteria:

* Diagnosis of secondary headache, based on clinical history, family history, neurological examination, or laboratory/imaging findings
* Failure to meet ICHD-3 diagnostic criteria for primary headache
* Presence of structural brain lesions or other neurological disorders
* Chronic systemic illness or current use of other migraine prophylactic medications
* Incomplete data or loss to follow-up within the 3-month period

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of pediatric patients aged [2-19] who were diagnosed with primary headache disorders, specifically migraine, according to the International Classification of Headache Disorders, 3rd edition (ICHD-3). Participants were evaluated and followed at the pediatric neurology outpatient clinic of a tertiary care hospital between January 2021 and December 2023. Patients with confirmed comorbid conditions (e.g., anxiety, benign paroxysmal vertigo, essential tremor) and/or vitamin deficiencies were included to assess the impact of these factors on treatment response. Those with secondary headache, neurological disorders, or incomplete records were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pediatric Migraine Disability Assessment Scale (PedMIDAS) Score | Baseline to 3 months after treatment
  The primary outcome is the change in PedMIDAS score from baseline to 3 months after treatment. PedMIDAS is a validated questionnaire that quantifies migraine-related disability in children and adolescents. A greater reduction indicates improved clinical response.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Scores | Baseline to 3 months after treatment
  VAS pain scores range from 0 (no pain) to 10 (worst imaginable pain). The change in VAS score after 3 months of treatment reflects the patient's subjective pain improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No